CLINICAL TRIAL: NCT06802250
Title: Effects of a Multi-component Early Child Development Intervention in Middle- Childhood: a Follow-up Study of the RINEW Randomized Controlled Trial
Brief Title: RINEW Randomized Controlled Trial 7-year Follow-up
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: Stanford University (Other); Purdue University (Other); International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024-02-17211
Record Dates: First submitted 2024-12-30; First posted 2025-01-31 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Child Development
Keywords: Child development; Water, Sanitation, and Hygiene; Nutrition; Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessment team is separate from the implementation team, and are not aware of intervention components. Materials provided in the intervention (books, toys) may be visible in the participants homes, but the outcome assessment team was not aware that these are related to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control arm (No Intervention): No intervention administered
- Group only arm (Experimental): Participants were encouraged to attend fortnightly courtyard group meetings
  Interventions: Behavioral: RINEW intervention
- Combined delivery arm (Experimental): Participants were visited by community health promoters once a month in their home as well as receive encouragement to attend monthly courtyard group meetings in between the monthly home visits.
  Interventions: Behavioral: RINEW intervention

INTERVENTIONS:
Behavioral: RINEW intervention — The intervention included behavioral recommendations and guidance on the topics of Nutrition, WASH, Lead exposure prevention, Mental Health, and child stimulation. The intervention also included the provision of nutritional supplements based on age and nutritional status, low-cost picture books and toys, and soapy water bottles.
  Arms: Combined delivery arm; Group only arm

SUMMARY:
This study is designed to evaluate the impact of the RINEW multicomponent early child development intervention on child development and risk factors for poor child development in middle childhood. This study is a follow-up assessment of the children and primary caregivers enrolled in the RINEW cluster randomized controlled trial approximately 6 years following intervention completion.

ELIGIBILITY:
Inclusion Criteria: Child's primary caregiver was enrolled in the RINEW cluster randomized trial

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 620 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Wechsler Intelligence Scale for Children: 5th Edition (WISC-V) | 6 years after intervention completion
  The WISC-V assessment measures cognitive development and general intellectual abilities in children 6 years 0 months to 16 years 11 months of age (6:0-16:11). Higher scores represent better outcomes.
Child Socioemotional Development | 6 years after intervention completion
  Maternal-report questionnaire designed to measure psychological adjustment in children and aims to detect any emotional or behavioural problems.
Self-regulation | 6 years after intervention completion
  Observation of children's self-regulation during the administration of the WISC-V assessment.
Academic Achievement | 6 years after intervention completion
  Direct assessments of children's reading and math performance

SECONDARY OUTCOMES:
Caregiver Mental Health | 6 years after intervention completion
  Center for Epidemiologic Studies Depression Scale (20 questions). Higher scores represent more depressive symptoms experienced.
Home Environment | 6 years after intervention completion
  The middle childhood Home Observation for Measurement of the Environment (HOME) includes both caregiver report and observational items to assess the quality and quantity of stimulation and support available to the child at home.
School Grade Level | 6 years after intervention completion
  Parental report of child's current (or previous if no longer in school) grade level.
Presence of Improved Latrine | 6 years after intervention completion
  Observation
Presence of Handwashing Station with Soap and Water | 6 years after intervention completion
  Observation
Knowledge of lead | 6 years after intervention completion
  Participant response to question "do you know what lead is?"
Bone Lead Levels | 6 years after intervention completion
  X-ray fluorescence analysis of micrograms of lead per gram bone material

OTHER OUTCOMES:
Knowledge of 7 factors related to children's intelligence | 6 years after intervention completion
  Record of mention of 7 factors in response to question "What are the things that affect a child's intelligence?". Factors are: clean environment, parental involvement, nutrition, learning/education at home, learning/education outside of the home, communication, social stimulation.
Knowledge of ways to avoid harm from lead | 6 years after intervention completion
  Correct response to question "What ways do you know to avoid harm from lead?"
Child screen time | 6 years after intervention completion
  Number of hours spent using a digital screen per week (on average, caregiver report)
Parental perceived intelligence | 6 years after intervention completion
  Parental rating of child's intelligence (1-7)

CONTACTS AND LOCATIONS:
Overall Officials: Lia Fernald, PhD, Principal Investigator — University of California, Berkeley
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data collected for this study will be available on request within 5 years following the completion of data collection.
Supporting Information: SAP
Time Frame: Within 5 years following the completion of data collection.
Access Criteria: Completion of a signed data-sharing agreement access agreement; use for research purposes only.